CLINICAL TRIAL: NCT05995314
Title: Effects Of Different Doses Of Caffeine On Cognitive Performance In Healthy Physically Active Individuals
Brief Title: Effects Of Caffeine On Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CAF_MR_2023
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Caffeine
Keywords: ergogenic aid; sport performance; reaction time; anticipation; attention; memory
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To achieve the blinded placebo situation, a researcher not associated with the study will be performed the blinding and prepared identical capsules containing placebo or the corresponding dose of caffeine. This researcher will be assigned an alphanumeric code to each trial to blind participants and investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLACEBO (Placebo Comparator): placebo (0 mg/kg of body mass of caffeine). The capsule will be filled with 3 mg/kg of body mass of cellulose.
  Interventions: Dietary Supplement: PLACEBO
- 3mg/kg (Experimental): 3 mg/kg of body mass of caffeine (99% caffeine, Bulkpowders, United Kingdom).
  Interventions: Dietary Supplement: 3 mg/kg of caffeine
- 6mg/kg (Experimental): 6 mg/kg of body mass of caffeine (99% caffeine, Bulkpowders, United Kingdom).
  Interventions: Dietary Supplement: 6 mg/kg of caffeine

INTERVENTIONS:
Dietary Supplement: PLACEBO — 3 mg/kg of cellulose (0 mg/kg of caffeine)
  Arms: PLACEBO
Dietary Supplement: 3 mg/kg of caffeine — Ingestion of 3 mg/kg of body mass of caffeine
  Arms: 3mg/kg
Dietary Supplement: 6 mg/kg of caffeine — Ingestion of 6 mg/kg of body mass of caffeine
  Arms: 6mg/kg

SUMMARY:
Caffeine is a potent central nervous system stimulant that increases the activity in the prefrontal cortex and can improve cognitive skills. An improvement in these cognitive skills can lead to further benefits in athletic performance. Therefore, it is necessary to clarify the dose-response of caffeine on cognitive performance.The aim of this research will be to determine the effects of different doses of caffeine on sport-related cognitive aspects.

DETAILED DESCRIPTION:
The investigators will require healthy, physically active young adults to complete three trials under the conditions: a) placebo, b) 3 mg/kg, or c) 6 mg/kg body mass of caffeine. In each trial, different cognitive abilities will be assessed using the following test batteries: reaction time (DynavisionTM D2), anticipation (Bassin Anticipation Timer), sustained attention (Go/No-Go and Eriksen Flanker Test) and memory tests. In addition, side effects and the perceived sensation index will be recorded 24 h after each test.

ELIGIBILITY:
Inclusion Criteria:

* Physically active individuals ( >150 min/week moderate physical activity or >75 min/week vigorous physical activity)
* Individuals without serious and undiagnosed health problems.

Exclusion Criteria:

* Individuals with color blindness.
* Regular caffeine consumers (>3 cups of coffee/day).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Reaction Time | 10 minutes
  Reaction time (in seconds) shall be assessed with the Dynavision™ D2 Visomotor Device using the "Reaction Time Test". In this test the fastest visual, motor and physical reaction time will be measured.
Anticipation | 5 minutes
  Visual acuity related to hand-eye coordination and anticipation will be assessed using the Bassin Anticipation Timer instrument. The best anticipation time (in seconds) of each condition (5, 10 and 15 mph) will be taken.
Sustained attention | 10 minutes
  The ability of maintaining the attention and inhibiting an appropriate response will be measured by "Go/No-Go Test" [fastest, slowest, and average response time (in seconds), and successful attempts (percentage; %)] and "Eriksen Flanker Test" [congruent and incongruent reaction time (in seconds)].
Memory | 20 minutes
  To study the modulation of memory storage processes, three 20-item word lists were created. Each word in the list will be presented for 5 s. This will be followed by a 100 s memory consolidation interval, after which there will be a 120 s period in which as many words as the participants can remember will be written down (First time). After 15 min, participants will perform a recall task (Second time) in which they will have to rewrite all the words they remember at that time.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Abián-Vicén, PhD, Study Director — University of Castilla-La Mancha
Locations (1):
- Performance and Sport Rehabilitation Laboratory, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-delaCruz M, Esteban-Garcia P, Abian P, Bravo-Sanchez A, Pinas-Bonilla I, Abian-Vicen J. Effects of different doses of caffeine on cognitive performance in healthy physically active individuals. Eur J Nutr. 2024 Dec;63(8):3025-3035. doi: 10.1007/s00394-024-03486-9. Epub 2024 Sep 4. PMID 39231871